CLINICAL TRIAL: NCT01501591
Title: Interaction Between Drug and Placebo Effect:Randomized Placebo Controlled Trials May Not be Accurate in Determining Drug Effect Size
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: RAC 2111001
Record Dates: First submitted 2011-12-25; First posted 2011-12-29 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2016-02

CONDITIONS: Placebo Effect; Placebo Drug Interaction
Keywords: Placebo effect; placebo drug interaction; placebo -controlled clinical trials
MeSH Terms: interventions — Hydroxyzine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hydroxyzine (Other): This group will receive a first generation H-1 receptor antagonist, hydroxyzine (25 mg) twice on two days; on one day described by the investigator as hydroxyzine and on the other day described by the investigator as placebo, in a randomized balanced crossover design.
  Interventions: Drug: Hydroxizine
- Placebo (Other): This group will receive a placebo twice on two days; on one day described by the investigator as hydroxyzine and on the other day described by the investigator as placebo, in a randomized balanced crossover design.
  Interventions: Other: Placebo
- Hydroxyzine/placebo (Other): This group will receive hydroxyzine and placebo in a randomized double-blind placebo-controled crossover design.
  Interventions: Drug: hydroxyzine/placebo

INTERVENTIONS:
Drug: Hydroxizine — 25 mg orally, one time on two different days, 72 hours apart
  Arms: Hydroxyzine
Other: Placebo — Matching placebo once on two different days, 72 hours apart.
  Arms: Placebo
Drug: hydroxyzine/placebo — 25 mg hydroxyzine or placebo once on two different days, 72 hours apart
  Arms: Hydroxyzine/placebo

SUMMARY:
The total effect of a medication is the sum of its drug effect, placebo effect (meaning response of placebo), and their possible interaction. Current interpretation of the results of clinical trials (the gold standard in evidence based medicine) assumes no such interaction. Using a novel cross-over balanced placebo design and caffeine as a model drug, the investigators have recently shown that a negative interaction does exist; suggesting that the size of drug effect as currently measured by clinical trials may not be accurate. Due to the novelty of the findings and their important clinical practice and research implications, they need to be confirmed using another drug; and the size of drug effect measured using the novel design need to be directly compared to that measured using conventional clinical trial design. The results of the study are expected to further our understanding of a widely used medical intervention, i.e., placebo, and help assess the appropriateness of randomized clinical trials in determining the size of drug effect.

DETAILED DESCRIPTION:
BACKGROUND:

The total effect of a medication is the sum of its drug effect, placebo effect (meaning response of placebo), and their possible interaction. Current interpretation of the results of clinical trials (the gold standard in evidence based medicine) assumes no such interaction. Using a novel cross-over balanced placebo design and caffeine as a model drug we have recently shown that a negative interaction does exist; suggesting that the size of drug effect as currently measured by clinical trials may not be accurate. Due to the novelty of the findings and their important clinical practice and research implications, they need to be confirmed using another drug; and the size of drug effect measured using the novel design need to be directly compared to that measured using conventional clinical trial design.

DESIGN:

A cross-over balanced placebo plus randomized placebo-controlled clinical trial design.

METHODS:

480 adults will be double-blindly randomized to three groups: first generation H-1 receptor antagonist- hydroxyzine (25 mg), placebo, or hydroxyzine+placebo group. The first two groups will receive the assigned intervention described by the investigators as hydroxyzine or placebo, in a randomized crossover design. The third group will receive hydroxyzine and placebo in a randomized double-blind placebo-controled crossover design. Group assignment will be concealed from volunteers and recruiters. Data collectors will be blinded to group assignment and intervention assignment. Volunteers will be partially deceived to the intervention assignment in the first two groups and blinded in the third group. The interventions to the third group will be also administered blindly. Serum hydroxyzine levels will be determined 3 hours post intervention from all volunteers to verify compliance and help maintain deception/blinding. The results of the study are expected to further our understanding of a widely used medical intervention, i.e., placebo, and help assess the appropriateness of randomized clinical trials in determining the size of drug effect.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to 50 years;
* Being healthy,
* Able to abstain from smoking and alcohol
* Medication-free for one week
* Able to reproducibly express oneself using a 100 mm visual analog scale (VAS).

Exclusion Criteria:

* clinically relevant deviation from normal health
* pregnancy or lactation
* hypersensitivity to hydroxyzine or related compounds

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 480 (Actual)
Dates: Start 2012-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Area-under-the-curve for drowsiness | seven hours
  Seven-hour-area-under-the-curve of drowsiness on 100 mm visual analog scales will be determined
Area-under-the-curve for dryness of the mouth | seven hours
  Seven-hour-area-under-the-curve of dryness of the mouth on 100 mm visual analog scales will be determined

SECONDARY OUTCOMES:
Mean percent of time of reporting drowsiness on a dichotomous scale. | seven hours
  Mean percent of time of reporting drowsiness on a dichotomous scale will also be determined.
Mean percent of time of reporting dryness of mouth | seven hours
  Mean percent of time of reporting dryness of mouth on a dichotomous scale will also be determined.

CONTACTS AND LOCATIONS:
Locations (1):
- King Faisal Specialist Hospital & research Center, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Hammami MM, Hammami S, Al-Swayeh R, Al-Gaai E, Farah FA, De Padua SJ. Drug*placebo interaction effect may bias clinical trials interpretation: hybrid balanced placebo and randomized placebo-controlled design. BMC Med Res Methodol. 2016 Nov 29;16(1):166. doi: 10.1186/s12874-016-0269-1. PMID 27899067